CLINICAL TRIAL: NCT03853525
Title: Safety and Efficacy Evaluation of the Use of Bepantol® Derma Spray After Laser Depilation in the Inguinal Region in Adult Women - 21 Days Use at Home
Brief Title: A Study to Gain Information How Well Dexpanthenol Dermal Spray Helps the Skin to Recover After Laser Hair Removal in the Groin and Intimate Area
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20506
Record Dates: First submitted 2019-02-15; First posted 2019-02-25 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Skin Recovery
Keywords: Dermal spray; Laser depilation; Skin hydration; Consumer satisfaction; Sensorial perception
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women_Inguinal side BAY207543 (Experimental): Adult women apply BAY207543 randomized to one side of the inguinal region and semisolid vaseline to the other side of the inguinal region after laser depilation. The side with BAY207543 is investigated.
  Interventions: Drug: BAY207543 (Bepanthol, Bepantol® Derma Spray); Other: Semisolid vaseline
- Women_Inguinal side Vaseline (Active Comparator): Adult women apply BAY207543 randomized to one side of the inguinal region and semisolid vaseline to the other side of the inguinal region after laser depilation. The side with vaseline is investigated.
  Interventions: Drug: BAY207543 (Bepanthol, Bepantol® Derma Spray); Other: Semisolid vaseline

INTERVENTIONS:
Drug: BAY207543 (Bepanthol, Bepantol® Derma Spray) — Product is applied to one side of the inguinal region.
Other: Semisolid vaseline — Product is applied to one side of the inguinal region.

SUMMARY:
In this study, researchers want to learn more about the effect of dexpanthenol dermal spray on skin recovery after a dermatological procedure for hair removal (laser depilation) in the groin and intimate area in adult women.

After the hair removal procedure, participants will return within 3 weeks for 3 visits to the study center to investigate the skin condition such as redness, irritation, softness of skin and possible side effects. Study participants will also be asked about their general acceptance of dexpanthenol dermal spray.

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy of the test product to aid skin recovery after lasering depilation in the intima and inguinal region.

Secondary objectives comprise clinical efficacy with respect to skin hydration, softness, vitality, appearance etc. and skin recovery, consumer judgement of product performance and acceptability, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Phototypes I and II according to the Fitzpatrick scale
* Participants willing to have a dermatological procedure (laser depilation) in the inguinal region to remove hairs in the region

Exclusion Criteria:

* Pathologies and/or skin injuries, such as psoriasis, sensitive skin, skin cancer, atopic dermatitis or other medical criteria to be considered at the time of evaluation
* Hyperpigmentations in the test area that interfere with the evaluation of possible reactions (vascular malformations, scars, increase of pilosity and large amount of nevi)
* Pathologies and/or active skin injuries (local and/or disseminated) in the evaluation area

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss by TEWL probe | Up to 23 days
  The transepidermal water loss (TEWL) is measured in g m2 h-1 with a Tewameter TM300.

SECONDARY OUTCOMES:
Skin properties of the participants | Up to 23 days
  Investigators assess various skin properties of the participants with a questionnaire (each scored from 1 to 5), resulting in an overall efficacy score from 9 to 45 (a higher score represents higher efficacy).
Treatment satisfaction | Up to 23 days
  Participants assess their treatment satisfaction with a questionnaire consisting of 13 items (each item is scored from 1-5) resulting in a score range of 13 to 65 (a higher score represents better treatment satisfaction).
Product evaluation | Up to 23 days
  Participants assess their sensorial perception of different product attributes (e.g. smell, absorption) with a questionnaire consisting of 6 items (each item is scored from 1-5) resulting in a score range from 6 to 30 (a higher score represents higher product satisfaction).
Number of adverse events by dermatological evaluation | Up to 23 days
Severity of adverse events by dermatological evaluation | Up to 23 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.